CLINICAL TRIAL: NCT03979716
Title: Exploration de l'Odorat en Imagerie Par Résonance Magnétique Fonctionnelle Chez Les Patients Atteints de Polypose Nasosinusienne
Brief Title: Smell Exploration in Patients With Nasal Polyposis : Study by Functional Magnetic Resonance Imaging
Acronym: ODORAT_IRMf
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, NGUYEN, Medical Doctor, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-A03215-50
Record Dates: First submitted 2019-05-23; First posted 2019-06-07 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Nasal Polyposis
MeSH Terms: conditions — Nasal Polyps | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anosmic patients (Experimental)
  Interventions: Device: fMRI
- Hyposmic patients (Experimental)
  Interventions: Device: fMRI
- Normosmic patients (Experimental)
  Interventions: Device: fMRI

INTERVENTIONS:
Device: fMRI — fMRI examination

SUMMARY:
Nasal polyposis (NP) is a disease affecting 4% of the population. This disease is frequently accompanied by olfactory disorders (41%-84% of patients) that affect patients' quality of life.

The aim of this study is to show brain activity differences in olfactory areas before and after surgery in each patient and between patient groups (normosmic, hyposmic and anosmic one) using functional Magnetic Resonance Imaging (fMRI). Brain activity will be measured by the intensity of brain signals and of the size of olfactory areas during olfactory stimulation before and after surgery. We suppose that fMRI could predict whether or not the patient will be able to recover smell after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nasal polyposis managed in the department of otorhinolaryngology and head and neck surgery of Nancy University Hospital,
* Adult Patients,
* Justifying a surgical treatment for nasal polyposis,
* Present hyposmia, anosmia or normosmia before surgery (confirmed by threshold and identification tests of the Sniffin' Stick kit),
* Affiliated with or beneficiary of a social security scheme,
* Having received complete information about the study and having signed an informed consent form.

Exclusion Criteria:

* General contraindications to Magnetic Resonance Imaging,
* Female of childbearing age without effective contraception,
* Persons referred in Articles L. 1121-5 to L. 1121-8 and L1122-2 of the Public Health Code,
* Qualitative sense of smell disorder (cacosmia, hyperosmia, phantosmia, parosmia),
* Smell disorders with neurological, post-traumatic, or neurodegenerative origin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-06-23 (Estimated); Study Completion 2021-06-23 (Estimated)

PRIMARY OUTCOMES:
Functional Brain activity | 6 months after the last inclusion
  Blood Oxygen Level Dependent (BOLD) measures in olfactory areas during calibrated olfactory stimuli in patients with NP whose olfactory function is clinically normal (normosmia), decreased (hyposmia) or absent (anosmia).

SECONDARY OUTCOMES:
Functional Brain activity | 6 months after the last inclusion
  Changes in Blood Oxygen Level Dependent (BOLD) measurements in olfactory areas during calibrated olfactory stimuli before and after NP surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Duc Trung NGUYEN, MD, PhD, MPH, Principal Investigator — University Hospital, Nancy, France
Locations (1):
- CHRU de Nancy, Nancy, France